CLINICAL TRIAL: NCT00100230
Title: Investigation of Effectiveness and Safety of High Dose Docosahexaenoic Acid (DHA) in X-Linked Retinitis Pigmentosa
Brief Title: DHA and X-Linked Retinitis Pigmentosa
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Retina Foundation of the Southwest (Other)
Collaborators: Foundation Fighting Blindness (Other); DSM Nutritional Products, Inc. (Industry)
Responsible Party: Principal Investigator, Dennis Hoffman, Senior Research Scientist (Retina Foundation of the Southwest), Retina Foundation of the Southwest
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2543; FD-R-002543; 5R01FD002543 (FDA); C-TX02-0704-0274 (Other Grant/Funding Number: Foundation Fighting Blindness)
Record Dates: First submitted 2004-12-27; First posted 2004-12-28 (Estimated); Results first posted 2015-03-17 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Retinitis Pigmentosa; X-linked Genetic Diseases
Keywords: retina; electroretinography; clinical trial; docosahexaenoic acid; omega-3 fatty acid; x-linked inheritance
MeSH Terms: conditions — Retinitis Pigmentosa; Genetic Diseases, X-Linked | interventions — Docosahexaenoic Acids; Fatty Acids, Omega-3

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1. (Experimental): Oral Docosahexaenoic acid, dosage based on body weight
  Interventions: Drug: docosahexaenoic acid OR corn/soy oil placebo
- 2 (Placebo Comparator): corn/soy oil placebo; oil not containing DHA...dosage based on body weight
  Interventions: Drug: docosahexaenoic acid OR corn/soy oil placebo

INTERVENTIONS:
Drug: docosahexaenoic acid OR corn/soy oil placebo — daily intake of DHA based on body weight or corn/soy oil placebo(oil not containing DHA; 4 year trial
  Other Names: DHA; omega-3 fatty acid; OR RANDOMIZED TO corn/soy oil placebo

SUMMARY:
Purpose:

Retinitis pigmentosa (RP) is characterized by progressive loss of visual function due to specific genetic mutations. This trial is focused on patients with one of the most severe forms of the disease, X-linked inherited RP (XLRP). This disease is characterized by early onset (typically loss of night vision as a child) followed by loss of peripheral vision as a teenager and young adult. There is no male-to-male transmission of the disease in the family.

There is no cure for RP and treatment options are limited. Two clinical trials have not found a benefit from nutritional supplementation with the long-chain polyunsaturated fatty acid, docosahexaenoic acid (DHA), at low daily doses although there is evidence that it slows disease progression in certain instances. In this clinical trial, we propose that a high dose nutritional DHA supplement will slow the loss of visual function and preserve usable vision in patients with XLRP.

This study is a 4-year placebo-controlled randomized clinical trial meaning that patients have a 50-50 chance of receiving placebo or experimental treatment. A total of 66 patients will be enrolled; 33 will receive placebo and 33 will receive the treatment. Entry criteria include diagnosis of XLRP by an ophthalmologist, age 7 to 32 years, male, sufficient visual function such that disease progression can be followed for the entire duration of the trial, and a willingness to visit the testing site (Dallas, TX) once a year.

Annual visual function testing includes ETDRS visual acuity, full-field and multifocal electroretinography (ERG), static peripheral visual fields, and fundus photography. Cone ERG function is the primary outcome measure.

Funding Source - FDA, Foundation Fighting Blindness, DSM Nutritionals

DETAILED DESCRIPTION:
Location & Contact Information:

Retina Foundation of the Southwest, 9600 N. Central Expressway, Suite 200, Dallas, TX 75231 Contact: Dr. D. Hoffman (dhoffman@retinafoundation.org) or Dr. D. Birch (dbirch@retinafoundation.org).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of RP by a retinal specialist
* Clinical diagnosis consistent with X-linked inheritance
* Enrolling minors and young adults (early onset of X-linked disease; ages 7 to 32)
* Measurable cone ERG responses --patients with less than 0.64 microvolt response to 31-Hz flicker will be excluded as they are more likely to become undetectable during the study
* Both eyes must meet entry criteria as both will be tested (i.e., no cataracts requiring surgery or retinal detachments).
* Media clarity sufficient for fundus photography
* Able to return to study site at yearly intervals
* Willing to supply blood samples at 6-month intervals
* Judiciously take the placebo or DHA supplement for the 4-year study duration
* Patient/parent/guardian understands and signs consent form.

Exclusion Criteria:

* Excessive fish consumption (e.g., cold water fish such as salmon, tuna, sardines) and/or fish oil supplementation (or other oil containing DHA)
* Baseline RBC-DHA levels showing evidence of supplementation (a typical level of RBC-DHA in normals is about 3.8%)
* Chronic metabolic disease that may interfere with fatty acid metabolism or require anti-coagulant medication

No ethnic or racial groups will be excluded.

Ages: 7 Years to 32 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 78 (Actual)
Dates: Start 2004-09; Primary Completion 2012-05 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis R. Hoffman, Ph.D., Principal Investigator — Retina Foundation of the Southwest
Locations (1):
- Retina Foundation of the Southwest, Dallas, Texas, United States

REFERENCES:
- [Result] Hoffman DR, Hughbanks-Wheaton DK, Pearson NS, Fish GE, Spencer R, Takacs A, Klein M, Locke KG, Birch DG. Four-year placebo-controlled trial of docosahexaenoic acid in X-linked retinitis pigmentosa (DHAX trial): a randomized clinical trial. JAMA Ophthalmol. 2014 Jul;132(7):866-73. doi: 10.1001/jamaophthalmol.2014.1634. PMID 24805262
- [Result] Hughbanks-Wheaton DK, Birch DG, Fish GE, Spencer R, Pearson NS, Takacs A, Hoffman DR. Safety assessment of docosahexaenoic acid in X-linked retinitis pigmentosa: the 4-year DHAX trial. Invest Ophthalmol Vis Sci. 2014 Jul 11;55(8):4958-66. doi: 10.1167/iovs.14-14437. PMID 25015354
- [Derived] Hoffman DR, Hughbanks-Wheaton DK, Spencer R, Fish GE, Pearson NS, Wang YZ, Klein M, Takacs A, Locke KG, Birch DG. Docosahexaenoic Acid Slows Visual Field Progression in X-Linked Retinitis Pigmentosa: Ancillary Outcomes of the DHAX Trial. Invest Ophthalmol Vis Sci. 2015 Oct;56(11):6646-53. doi: 10.1167/iovs.15-17786. PMID 26469750
- [Derived] Cai CX, Locke KG, Ramachandran R, Birch DG, Hood DC. A comparison of progressive loss of the ellipsoid zone (EZ) band in autosomal dominant and x-linked retinitis pigmentosa. Invest Ophthalmol Vis Sci. 2014 Oct 23;55(11):7417-22. doi: 10.1167/iovs.14-15013. PMID 25342618
- [Derived] Birch DG, Locke KG, Wen Y, Locke KI, Hoffman DR, Hood DC. Spectral-domain optical coherence tomography measures of outer segment layer progression in patients with X-linked retinitis pigmentosa. JAMA Ophthalmol. 2013 Sep;131(9):1143-50. doi: 10.1001/jamaophthalmol.2013.4160. PMID 23828615
- See also: website for Retina Foundation of the Southwest — http://www.retinafoundation.org

RESULTS

PARTICIPANT FLOW:
Groups:
- 1. Docosahexaenoic Acid (DHA) Arm: Docosahexaenoic acid (an omega-3 polyunsaturated fatty acid) taken orally at a dosage of 30 mg/kg body weight/day for a 4-year duration trial.
- Corn/Soy Oil Placebo Arm: Corn/soy oil placebo (oils not containing DHA); dosage based on body weight for 4-year trial
Period: Overall Study
Arm/Group | 1. Docosahexaenoic Acid (DHA) Arm | Corn/Soy Oil Placebo Arm
Started | 41 | 37
Completed | 29 | 22
Not Completed | 12 | 15

BASELINE CHARACTERISTICS:
Population: males with X-linked retinitis pigmentosa
Groups:
- Total: Total of all reporting groups
Arm/Group | 1. Docosahexaenoic Acid (DHA) Arm | Corn/Soy Oil Placebo Arm | Total
Number analyzed (Participants) | 41 | 37 | 78
Age, Customized [Mean (Standard Deviation); unit: years] — Ages 7 to 32 years
  years
    Age | 16.7 (7.8) | 16.2 (6.6) | 16.7 (7.1)
Sex/Gender, Customized [Number; unit: participants]
  male | 41 | 37 | 78
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 37 | 33 | 70
  More than one race | 3 | 4 | 7
  Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 1 | 5
  Not Hispanic or Latino | 37 | 36 | 73
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 38 | 35 | 73
  Canada | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Rate of LOSS of 31 Hertz Cone Electroretinographic Function
Description: Hypothesis #1: Elevation of red blood cell-docosahexaenoic acid levels will slow the progressive loss of 31 hertz cone electroretinographic response in this 4-year trial.
Time Frame: 4 years
Population: Number of participants completing at least one year of trial (i.e., modified intent to treat cohort)
Measure: Mean (Standard Error); unit: log microvolts/year
Groups:
- DHA (Docosahexaenoic Acid): Oral Docosahexaenoic acid, dosage based on body weight
  docosahexaenoic acid OR corn/soy oil placebo: daily intake of DHA based on body weight or corn/soy oil placebo(oil not containing DHA; 4 year trial
- Placebo (Corn/Soy Oil): corn/soy oil placebo; oil not containing DHA...dosage based on body weight
  docosahexaenoic acid OR corn/soy oil placebo: daily intake of DHA based on body weight or corn/soy oil placebo(oil not containing DHA; 4 year trial
Arm/Group | DHA (Docosahexaenoic Acid) | Placebo (Corn/Soy Oil)
Number analyzed (Participants) | 33 | 27
log microvolts/year | 0.028 (0.001) | 0.022 (0.002)
Statistical Analysis 1: Comparison: DHA (Docosahexaenoic Acid) vs Placebo (Corn/Soy Oil); Test type: Non-Inferiority or Equivalence — Equivalence analysis: standard power calculation of 20%; used 2-sided t-test; p = 0.30, Mixed Models Analysis — Threshold for significance: p<0.05

2. Secondary Outcome: Rate of LOSS of Rod Electroretinographic Function
Description: Hypothesis #1: Elevation of red blood cell-docosahexaenoic acid levels will slow the progressive loss of rod electroretinographic response in this 4-year trial.
Time Frame: 4 years
Population: Number of participants completing at least one year of trial (i.e., modified intent to treat cohort)
Measure: Mean (Standard Error); unit: change in amplitude, log microvolts/year
Arm/Group | DHA (Docosahexaenoic Acid) | Placebo (Corn/Soy Oil)
Number analyzed (Participants) | 33 | 27
change in amplitude, log microvolts/year | 0.010 (0.001) | 0.023 (0.001)
Statistical Analysis 1: Comparison: DHA (Docosahexaenoic Acid) vs Placebo (Corn/Soy Oil); Test type: Non-Inferiority or Equivalence — Equivalence analysis: standard power calculation of 20%; used 2-sided t-test; p = 0.27, Mixed Models Analysis — Threshold for significance: p<0.05
Statistical Analysis 2: Comparison: DHA (Docosahexaenoic Acid) vs Placebo (Corn/Soy Oil); Test type: Non-Inferiority or Equivalence — Equivalence analysis: standard power calculation of 20%; used 2-sided t-test; p = 0.27, Mixed Models Analysis

3. Other Pre Specified Outcome: Loss of Peripheral Visual Fields
Description: Hypothesis: Elevation of red blood cell-docosahexaenoic acid levels will slow the progressive loss of peripheral visual fields in this 4-year trial.
Time Frame: 4 years
Population: Only participants completing at least one year of trial
Measure: Mean (Standard Error); unit: decibels (dB)
Groups:
- DHA (Docosahexaenoic Acid) ARM: Oral Docosahexaenoic acid, dosage based on body weight
  docosahexaenoic acid OR corn/soy oil placebo: daily intake of DHA based on body weight or corn/soy oil placebo(oil not containing DHA; 4 year trial
- Placebo (Corn/Soy Oil) ARM: corn/soy oil placebo; oil not containing DHA...dosage based on body weight
  docosahexaenoic acid OR corn/soy oil placebo: daily intake of DHA based on body weight or corn/soy oil placebo(oil not containing DHA; 4 year trial
Arm/Group | DHA (Docosahexaenoic Acid) ARM | Placebo (Corn/Soy Oil) ARM
Number analyzed (Participants) | 33 | 27
decibels (dB) | 50.4 (3.2) | 112.8 (2.0)
Statistical Analysis 1: Comparison: DHA (Docosahexaenoic Acid) ARM vs Placebo (Corn/Soy Oil) ARM; Test type: Non-Inferiority or Equivalence — Equivalence analysis: standard power calculation of 20%; used 2-sided t-test; p = 0.000008, Mixed Models Analysis — Threshold for significance: p<0.05

ADVERSE EVENTS:
Time Frame: 4 years
Description: Adverse events criteria were based on: Division of AIDS (DAIDS) National Institutes of Health. Table for grading severity of adult and pediatric adverse events (Dec 2004; rev. 2009) (http://rsc.tech-res.com/Document/safetyandpharmacovigilance/Table_for_Grading_Severity_of_Adult_Pediatric_Adverse_Events.pdf). Date of last access: 3-19-2014.
Arm/Group | 1. Docosahexaenoic Acid (DHA) Arm | Corn/Soy Oil Placebo Arm
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/27
Other Adverse Events (participants affected / at risk) | 9/33 | 16/27
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1. Docosahexaenoic Acid (DHA) Arm (N=33) | Corn/Soy Oil Placebo Arm (N=27)
Stomach ache (Gastrointestinal disorders) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (3)
Low HDL cholesterol (Blood and lymphatic system disorders) | 2 (2) | 5 (5)
elevated LDL cholesterol (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
elevated total cholesterol (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
elevated potassium (Blood and lymphatic system disorders) | 0 (0) | 4 (4)
elevated glucose (Blood and lymphatic system disorders) | 0 (0) | 3 (3)

LIMITATIONS AND CAVEATS:
A lower than expected event rate for the primary outcome measure was the major trial limitation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No